CLINICAL TRIAL: NCT02605577
Title: Research of Systemic Management for Late Preterm Infants Nutrition in China
Acronym: NLP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University First Hospital (Other); Peking University People's Hospital (Other); Peking University Third Hospital (Other); Beijing Children's Hospital (Other); Capital Institute of Pediatrics, China (Other); Beijing Obstetrics and Gynecology Hospital (Other); Beijing Huaxin Hospital (Unknown); Beijing Friendship Hospital (Other); Beijing Ditan Hospital (Other); Bayi Children's Hospital Affiliated to Beijing Military Gen Hospital (Unknown); Beijing Shangdi Hospital (Unknown); Beijing Tongzhou District Maternal and Child Health Hospital (Unknown); Beijing Yanqing County Hospital (Unknown); People's Hospital of Beijing Daxing District (Other); Beijing Hospital (Other Government); Civil Aviation General Hospital (Other); Beijing Anzhen Hospital (Other); Military 301 Hospital (Unknown); Beijing Haidian Maternal and Child Health Hospital (Other); Beijing 302 Hospital (Other); Beijing Chaoyang District Maternal and Child Health Hospital (Unknown); China-Japan Friendship Hospital (Other); Military 306 Hospital (Unknown); Beijing Chao Yang Hospital (Other); Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Li zhenghong, associate professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMFLPIN
Record Dates: First submitted 2015-10-06; First posted 2015-11-16 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Late Premature Infants; Systemic Nutritional Management
Keywords: late preterm infants; nutrition; systemic management

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (Experimental): group of late preterm infants following "new systemic nutritional management protocol" during hospital stay,which including specific enteral and parenteral nutritional protocol and complication monitor, such as hyperglycemia,hypoglycemia,infection,hyperbilirubinemia and anemia(the intervention refers to this"new systemic nutritional management protocol" )
  Interventions: Procedure: new systemic nutrition management protocol
- control group (No Intervention): group of late preterm infants using current nutritional management protocol during hospital stay

INTERVENTIONS:
Procedure: new systemic nutrition management protocol — a new established systemic nutrition management protocol
  Arms: experimental group

SUMMARY:
The purpose of the project is to investigate the status of nutrition management of late preterm infants in the member hospitals in the Beijing association of preterm infants, and set up the systemic nutritional management of late preterm infants, Including parenteral nutrition and enteral feeding. And to compare the differences of growth and complications of these infants between groupings applicationg and not applicating the systemic nutritional management of late preterm infants,and to validate its feasibility and validity.

DETAILED DESCRIPTION:
The research content of the project includes three parts:

1. Investigation on nutritional status of late preterm infants.
2. Setting up systemic nutritional management of late preterm infants
3. Comparing nutritional and growth status of the late preterm, short-term and long-term complications between the groups applicating and not applicating the systemic nutritional management of late pretern infants.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants with gestational age 34 weeks to 36 weeks and 6 days

Exclusion Criteria:

* preterm infants with gestational age<34 weeks or >36 weeks and 6 days
* abnormality of digestive system
* genetic and metablic disease
* severe congenital heart disease( with hemodynamic changes that influencing enteral feeding)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
days of postnatal life when enteral nutrition reaching 120kcal/kg/d | 29 months
weight gain(g/kg/week) | 29 months
length gain(cm/week) | 29 months
circumference gain(cm/week) | 29 months

SECONDARY OUTCOMES:
days of postnatal life when reaching full enteral nutrion(d) | 29 months
  the incidence of complications of preterm infants
proportion of breast milk feeding(%) | 29 months
days of postnatal life with the lowst weight during hospitalisation(d) | 29 months
the lowest weight during hospitalisation(g) | 29 months
days of postnatal life that regain birth weight(d) | 29 months
incidence of hyperglycemia(%) | 29 months
incidence of hypoglycemia(%) | 29 months
incidence of hypebilirubinemia(%) | 29 months
incidence of neonatal infection(%) | 29 months
incidence of neonatal anemia(%) | 29 months